CLINICAL TRIAL: NCT07062731
Title: Effect of Pelvic Floor Muscle Exercises on Women With Suboptimal Anorectal Manometry Results After an Obstetric Anal Sphincter Injury (OASI)
Brief Title: Pelvic Floor Exercises for Suboptimal Anorectal Manometry
Status: Recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Kar Yee Lor, Dr. Kar Yee Lor, King's College Hospital NHS Trust
Other Study IDs: IRAS 353671
Record Dates: First submitted 2025-06-26; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Obstetric Anal Sphincter Injury
Keywords: pelvic floor muscle exercises

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obstetric anal sphincter injury (suboptimal/ abnormal): Women who have sustained an obstetric anal sphincter injury and was found to have suboptimal (20-40mmHg) or abnormal (<20mmHg) incremental squeeze pressure on anorectal manometry
  Interventions: Behavioral: Supervised pelvic floor muscle exercises

INTERVENTIONS:
Behavioral: Supervised pelvic floor muscle exercises — 4 months of supervised physiotherapy by a women's health physiotherapists (3 sessions in total)

SUMMARY:
Currently, guidelines from the Royal College of Obstetricians and Gynaecologists stipulate that all women who have sustained an obstetric anal sphincter injury in a previous pregnancy and who are symptomatic or have abnormal endoanal ultrasonography and/ or manometry should be counselled regarding the option of an elective Caesarean section. An abnormal endoanal ultrasonography is currently considered to be a defect of the external anal sphincter (EAS) of more than 30 degrees while an abnormal anorectal manometry would be an incremental squeeze pressure of less than 20mmHg.

This study aims to evaluate if a course of guided pelvic floor exercises could improve anal sphincter function on those with suboptimal or abnormal anal incremental squeeze pressures, and subsequently expand their options for future modes of delivery (vaginal delivery not contraindicated)

ELIGIBILITY:
Inclusion Criteria:

1. Female patients who have sustained an obstetric anal sphincter injury after their most recent delivery and:

   1. Are at least 6 weeks postpartum
   2. Has not received any form of guided pelvic floor exercises by a licensed women's health physiotherapist postpartum
2. Either able to speak, read and write in English, or has a professional interpreter present at the time of appointment.
3. Capable of understanding and signing the informed consent form after full discussion of the investigations and its risks and benefits.
4. Able and willing to complete the St Mark's Score, ICIQ-UI SF and other trial related questionnaires, comply with scheduled clinic visits and manometry studies.

Exclusion Criteria:

* Inclusion Criteria

  1. Female patients who have sustained an obstetric anal sphincter injury after their most recent delivery and:

     1. Are at least 6 weeks postpartum
     2. Has not received any form of guided pelvic floor exercises by a licensed women's health physiotherapist postpartum
  2. Either able to speak, read and write in English, or has a professional interpreter present at the time of appointment.
  3. Capable of understanding and signing the informed consent form after full discussion of the investigations and its risks and benefits.
  4. Able and willing to complete the St Mark's Score, ICIQ-UI SF and other trial related questionnaires, comply with scheduled clinic visits and manometry studies.

Exclusion Criteria

1. Women who have sustained an obstetric anal sphincter injury more than a year ago
2. Women who have had another vaginal delivery after sustaining an obstetric anal sphincter injury in a previous delivery.
3. Existing anal pain precluding anorectal examination
4. Existing neurological, musculoskeletal disorders which impedes ability to perform pelvic floor muscle exercises
5. Age <18 years old
6. Currently pregnant
7. Inability to comply with pelvic floor muscle exercises

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women who have delivered at either Kings College Hospital or Princess Royal Hospital, have sustained an obstetric anal sphincter injury and have suboptimal or abnormal incremental squeeze pressures during anorectal manometry at perineal clinic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Success | 4 months
  1. Change of incremental squeeze pressure from abnormal (<20mmHg) or suboptimal (20-40mmHg) to normal (>40mmHg)
  2. Change of incremental squeeze pressure from abnormal (<20mmHg) to suboptimal (20-40mmHg)

SECONDARY OUTCOMES:
Change or recommended mode of delivery | 4 months
  Change of recommended mode of delivery from elective Caesarean section only to spontaneous vaginal delivery or elective Caesarean section
Change in St Mark's Score | 4 months
  Change in St Mark's score before and after intervention
Change in International Consultation on Incontinence Questionnaire- Urinary Incontinence Short Form (ICIQ-UI SF) | 4 months
  Change in ICIQ-UI SF before and after intervention
Change in Faecal Incontinence Quality of life Scale | 4 months
  Change in Faecal Incontinence Quality of life Scale before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Kings College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No